CLINICAL TRIAL: NCT02037438
Title: Sustainable Methods, Algorithms, and Research Tools for Delivering Optimal Care Study (SMART DOCS)
Brief Title: Sustainable Methods, Algorithms, and Research Tools for Delivering Optimal Care Study
Acronym: SMART DOCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Clete A. Kushida, Principle Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CE-12-11-4137; SPO #: 105981 (Other: Stanford Sponsored Project Number)
Record Dates: First submitted 2014-01-14; First posted 2014-01-16 (Estimated); Results first posted 2019-03-04 (Actual); Last update posted 2019-03-04 (Actual); Status verified 2018-11

CONDITIONS: Obstructive Sleep Apnea of Adult; Insomnia; Circadian Rhythm Sleep Disorder; Sleep Related Movement Disorders; Narcolepsy and Hypersomnia; Parasomnia
Keywords: Clinical sleep medicine; New methodology for healthcare delivery; Diagnosis and treatment of sleep disorders; Electronic health records; Clinical informatics; Evidence-based comparative effectiveness research; Sleep specialists; Primary care providers; Allied health professionals; Patient-centered care
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Disorders, Circadian Rhythm; Narcolepsy; Disorders of Excessive Somnolence; Parasomnias; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CONV Arm (Active Comparator): Conventional (CONV) care for the diagnosis and treatment of sleep disorders
  Interventions: Other: CONV care for the diagnosis and treatment of sleep disorders
- PCCM ARM (Experimental): Patient-Centered Outcomes and Coordinated Care Management (PCCM) for the diagnosis and treatment of sleep disorders
  Interventions: Other: PCCM for the diagnosis and treatment of sleep disorders

INTERVENTIONS:
Other: CONV care for the diagnosis and treatment of sleep disorders — The Conventional (CONV) intervention utilized standard-of-care diagnostic and treatment procedures for new patients with sleep disorders at the Stanford Sleep Medicine Center
  Arms: CONV Arm
Other: PCCM for the diagnosis and treatment of sleep disorders — The Patient-Centered Outcomes and Coordinated Care Management (PCCM) intervention implemented new methodologies for the diagnosis and treatment of sleep disorders. It also incorporates the utilization of a web-based interactive portal that provides specific and relevant information and resources for patients, health care providers, and allied health professionals. The portal was designed to facilitate informed health care decisions among patients and health care providers through improved access to medical data and enhanced communications.
  Arms: PCCM ARM

SUMMARY:
Sustainable Methods, Algorithms, and Research Tools for Delivering Optimal Care Study (SMART DOCS) was designed to develop and evaluate a new approach (patient-centered outcomes and coordinated-care management [PCCM]) for the diagnosis and treatment of sleep disorders. Specialized and pertinent information and resources regarding sleep disorder management were developed and made available through an online portal, allowing patients to make informed health care decisions, and providers to assist patients in achieving what they feel are the most important goals regarding their care. Half of participants were randomized into the conventional diagnosis and treatment (CONV) arm and the other half into the patient-centered outcomes and coordinated-care management (PCCM) arm. Validated objective and subjective assessment measures were administered at intervals throughout a 13 month participation period in both the CONV and PCCM arms to determine whether the new PCCM approach for sleep medicine results in increased patient satisfaction, quality of care, and improved health outcomes. Qualifying participants were 18 years of age or older and presenting with a new sleep disorder. Patients received no monetary compensation.

DETAILED DESCRIPTION:
SMART DOCS is a randomized comparative clinical trial designed to evaluate a new approach of outpatient medical care. In current sleep medicine practice, a consultation lasting one hour or less is allotted for the assessment, diagnosis, planning, and implementation of sleep disorders among patients and their health care provider. Patients are expected to convey their complex medical history and relevant symptoms, while clinicians must effectively and appropriately diagnose and create a treatment plan in this given period of time.

New technology for home-based diagnostic testing and electronic access to diagnostic results and outcomes provides functional advantages to the delivery of healthcare in an outpatient setting. The project was designed to compare the traditional diagnostic and treatment medical outpatient approach to a patient-centered outcomes and coordinated-care management (PCCM) approach for sleep medicine. New or refined methods, algorithms, and tools were expected to improve clinical practice and the patient's experience of care. The specific aim of this study was to determine whether a new patient-centered outcomes and coordinated-care management (PCCM) approach for sleep medicine provides better care and improves the health of patients compared to a conventional diagnostic/treatment outpatient medical care (CONV) approach.

Patients were randomized to one of two arms; Conventional Diagnostic/Treatment Outpatient Medical Care (CONV) and Patient-Centered Outcomes and Coordinated-Care Management (PCCM). Randomization was conducted using a permuted block design. Each new patient consecutively seen at the Stanford Sleep Medicine Center and each patient seen at Stanford Sleep Clinic in Primary Care who were suspected of having a new sleep disorder were informed about the study. The patient was notified that the study was a randomized trial and he or she could be assigned to either the CONV or PCCM arms. The patient was also apprised that he or she was consenting to grant access all clinical data collected during his or her evaluation and treatment to the research team. If the patient agreed to participate, informed consent was obtained. He or she was then randomized to one of the study arms in order to diagnose and treat his or her sleep disorder.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* New clinical outpatient presenting signs and/or symptoms of a sleep disorder

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1836 (Actual)
Dates: Start 2014-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clete A Kushida, M.D., Ph.D., Principal Investigator — Stanford University
Locations (1):
- Stanford Sleep Clinic, Stanford University Center for Sleep Science and Medicine, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with other researchers; these data will be available after April 2017

REFERENCES:
- [Background] Kushida CA, Nichols DA, Holmes TH, Miller R, Griffin K, Cardell CY, Hyde PR, Cohen E, Manber R, Walsh JK. SMART DOCS: a new patient-centered outcomes and coordinated-care management approach for the future practice of sleep medicine. Sleep. 2015 Feb 1;38(2):315-26. doi: 10.5665/sleep.4422. PMID 25409112

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CONV Arm | PCCM ARM
Started | 920 | 916
Completed | 574 | 561
Not Completed | 346 | 355

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CONV Arm | PCCM ARM | Total
Number analyzed (Participants) | 920 | 916 | 1836
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.1 (15.60) | 49.1 (14.98) | 50.1 (15.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 396 | 401 | 797
  Male | 524 | 515 | 1039
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 89 | 97 | 186
  Not Hispanic or Latino | 814 | 808 | 1622
  Unknown or Not Reported | 17 | 11 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 11 | 8 | 19
  Asian | 146 | 103 | 249
  Native Hawaiian or Other Pacific Islander | 8 | 8 | 16
  Black or African American | 32 | 23 | 55
  White | 607 | 677 | 1284
  More than one race | 105 | 88 | 193
  Unknown or Not Reported | 11 | 9 | 20
Region of Enrollment [Number; unit: participants]
  United States | 920 | 916 | 1836

OUTCOME MEASURES:

1. Primary Outcome: Change in CGCAHPS Global Rating After 12 Months
Description: Global rating of the provider from the Consumer Assessment of Healthcare Providers and Systems Clinician and Group Survey (CGCAHPS) compared between the two arms at end of study (12 months). The global rating instructions specify: "Using any number from 0 to 10, where 0 is the worst provider possible, and 10 is the best provider possible, what number would you use to rate this provider?"
Time Frame: 12 months
Population: Although 1135 participants (574 CONV, 561 PCCM) completed at least one of the primary outcome measures, 546 CONV and 535 PCCM participant data were acceptable for statistical analysis for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CONV Arm | PCCM ARM
Number analyzed (Participants) | 546 | 535
units on a scale | 8.32 (1.973) | 8.45 (1.650)
Statistical Analysis 1: Comparison: CONV Arm vs PCCM ARM; Test type: Superiority or Other; p = 0.687, see Comments; Finite-Mixture Models with Fixed Effects for Providers; Provider-Effect Adjusted Difference = 0.03, Standard Error of Mean 0.075

2. Primary Outcome: Change in SF-36 Version 2 Health Survey Vitality Score After 12 Months
Description: The vitality scale score of the Short Form-36 (SF-36) Version 2 Health Survey was compared at the end-of study (12 months) and was derived from the following four questions: "How much of the time during the past 4 weeks… Did you feel full of life?" "Did you have a lot of energy?" "Did you feel worn out?" "Did you feel tired?" The possible responses and point values were: all of the time (1), most of the time (2), some of the time (3), a little of the time (4), and none of the time (5). The scale is transformed to a 0-100 scale, with the lower the score indicating more disability.
Time Frame: 12 months
Population: Although 1135 participants (574 CONV, 561 PCCM) completed at least one of the primary outcome measures, 540 CONV and 539 PCCM participant data were acceptable for statistical analysis for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CONV Arm | PCCM ARM
Number analyzed (Participants) | 540 | 539
units on a scale | 48.0 (10.84) | 47.1 (11.19)
Statistical Analysis 1: Comparison: CONV Arm vs PCCM ARM; Test type: Superiority or Other; p = 0.989, see Comments; Heteroscedasticity-Consistent Linear Regression with Fixed Effects for Providers and Baseline Covariate; Provider-Effect Adjusted Difference = -0.007, Standard Error of Mean 0.539

3. Secondary Outcome: Change in CGCAHPS Provider Communication After 12 Months
Description: Communication of provider as measured by the Consumer Assessment of Healthcare Providers and Systems Clinician and Group Survey (CGCAHPS). This comprised "How Well Providers (or Doctors) Communicate with Patients" The ratings for the following four questions were averaged for each participant: "In the last 12 months, how often did this provider explain things in a way that was easy to understand?" "In the last 12 months, how often did this provider listen carefully to you?" "In the last 12 months, how often did this provider show respect for what you had to say?" "In the last 12 months, how often did this provider spend enough time with you?" The responses and point values were: never (1), sometimes (2), usually (3), and always (4).
Time Frame: 12 months
Population: Although 1135 participants (574 CONV, 561 PCCM) completed at least one of the primary outcome measures, 530 CONV and 525 PCCM participant data were acceptable for statistical analysis for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CONV Arm | PCCM ARM
Number analyzed (Participants) | 530 | 525
units on a scale | 3.59 (0.655) | 3.64 (0.551)
Statistical Analysis 1: Comparison: CONV Arm vs PCCM ARM; Test type: Superiority or Other; p = 0.417, see Comments; Finite-Mixture Models with Fixed Effects for Providers; Provider-Effect Adjusted Difference = 0.114, Standard Error of Mean 0.141

4. Secondary Outcome: Change in CGCAHPS Health Information Technology Measure #1 After 12 Months
Description: Helpfulness of Provider's Use of Computers During a Visit (Effectiveness of technology as measured by the Health Information Technology item set of the Consumer Assessment of Healthcare Providers and Systems Clinician and Group Survey [CGCAHPS]). This included composite measures of helpfulness of provider's use of computers during a visit. The ratings for the following two questions were averaged for each participant: "During your visits in the last 12 months, was this provider's use of a computer or handheld device helpful to you?" The point values for the responses were: yes, definitely (1), yes, somewhat (2), and no (3). "During your visits in the last 12 months, did this provider's use of a computer or handheld device make it harder or easier for you to talk with him or her?" The point values for the responses were: easier (1), not harder or easier (2), harder (3).
Time Frame: 12 months
Population: Although 1135 participants (574 CONV, 561 PCCM) completed at least one of the primary outcome measures, 423 CONV and 426 PCCM participant data were acceptable for statistical analysis for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CONV Arm | PCCM ARM
Number analyzed (Participants) | 423 | 426
units on a scale | 2.03 (0.378) | 2.06 (0.356)
Statistical Analysis 1: Comparison: CONV Arm vs PCCM ARM; Test type: Superiority or Other; p = 0.468, see Comments; Finite-Mixture Models with Fixed Effects for Providers; Provider-Effect Adjusted Difference = 0.057, Standard Error of Mean 0.078

5. Secondary Outcome: Change in CGCAHPS Health Information Technology Measure #3 After 12 Months
Description: Helpfulness of Provider's Website in Giving Patient Information About Patient's Care and Tests (Effectiveness of technology as measured by the Health Information Technology item set of the Consumer Assessment of Healthcare Providers and Systems Clinician and Group Survey [CGCAHPS]). This included composite measures of helpfulness of provider's website in giving information about care and tests. The ratings for the following four questions were averaged for each participant: "In the last 12 months, how often was it easy to find these lab or other test results on the website?" "In the last 12 months, how often were these lab or other test results put on the website as soon as you needed them?" "In the last 12 months, how often were these lab or other test results presented in a way that was easy to understand?" "In the last 12 months, how often were the visit notes easy to understand?" The responses and point values were: never (1), sometimes (2), usually (3), and always (4).
Time Frame: 12 months
Population: Although 1135 participants (574 CONV, 561 PCCM) completed at least one of the primary outcome measures, 268 CONV and 270 PCCM participant data were acceptable for statistical analysis for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CONV Arm | PCCM ARM
Number analyzed (Participants) | 268 | 270
units on a scale | 3.31 (0.787) | 3.30 (0.771)
Statistical Analysis 1: Comparison: CONV Arm vs PCCM ARM; Test type: Superiority or Other; p = 0.003, see Comments; Finite-Mixture Models with Fixed Effects for Providers; Provider-Effect Adjusted Difference = 0.177, Standard Error of Mean 0.061

ADVERSE EVENTS:
Time Frame: 1 year
Description: Only a subset of the total enrolled patients could be tracked for Serious Adverse Events. Other (Not Including Serious) Adverse Events were not recorded in the study. Serious Adverse Events were grouped into major organ system categories decided upon by the research team.
Arm/Group | CONV Arm | PCCM ARM
Serious Adverse Events (participants affected / at risk) | 30/158 | 23/172
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CONV Arm (N=158) | PCCM ARM (N=172)
Emergency Department Visits (Gastrointestinal disorders) | 1 | 0
Emergency Department Visits (Renal and urinary disorders) | 1 | 0
Emergency Department Visits (General disorders) | 0 | 1
Emergency Department Visits (Musculoskeletal and connective tissue disorders) | 0 | 1
Emergency Department Visits (Nervous system disorders) | 1 | 1
Emergency Department Visits (Psychiatric disorders) | 1 | 0
Hospital Admissions (Cardiac disorders) | 1 | 0
Hospital Admissions (Skin and subcutaneous tissue disorders) | 0 | 1
Hospital Admissions (Gastrointestinal disorders) | 0 | 1
Hospital Admissions (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hospital Admissions (Nervous system disorders) | 2 | 0
Hospital Admissions (Psychiatric disorders) | 1 | 0
Surgeries/Procedures (Cardiac disorders) | 3 | 4
Surgeries/Procedures (Endocrine disorders) | 1 | 0
Surgeries/Procedures (Gastrointestinal disorders) | 1 | 3
Surgeries/Procedures (Renal and urinary disorders) | 1 | 2
Surgeries/Procedures (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Surgeries/Procedures (General disorders) | 0 | 2
Surgeries/Procedures (Musculoskeletal and connective tissue disorders) | 4 | 4
Accidents (Musculoskeletal and connective tissue disorders) | 2 | 1
Deaths (Cardiac disorders) | 2 | 0
Deaths (Endocrine disorders) | 1 | 0
Deaths (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deaths (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No